CLINICAL TRIAL: NCT00473577
Title: Two Phase, Open-Label, Sequential, Ascending Dose Study of the Tolerability, Safety, and Pharmacokinetics of CRA-024781 in Cancer Patients
Brief Title: Study of the Tolerability, Safety, and Pharmacokinetics of CRA-024781 in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC 0401
Record Dates: First submitted 2007-05-11; First posted 2007-05-15 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Hematologic Neoplasms; Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CRA-24781

SUMMARY:
To determine the maximum tolerated dose (MTD) of CRA-024781 IV given by 2-hour intravenous infusions in patients with refractory solid or hematologic malignancies. To evaluate safety and tolerability, pharmacokinetics and pharmacodynamics, and to evaluate bioavailability of CRA-024781 IV when administered in a single oral dose.

DETAILED DESCRIPTION:
Patients will receive a single oral dose of CRA-024781 one week before beginning intravenous dosing. Blood samples for pharmacokinetic and pharmacodynamic analysis will be collected on several occasions prior to the start of the intravenous treatment.

The intravenous treatment will consist of 3 consecutive days of CRA-024781 IV administered as a 2-hour IV infusion every 3 weeks in a 4 weeks cycle.

Assessment of the extent of disease will be performed every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* histologically confirmed solid or hematologic malignancy that is refractory to standard therapy or for which no standard therapy exists
* estimated life expectancy > 12 weeks
* ECOG performance grade ≤ 2
* creatinine ≤ 1.5 X institutional upper limit of normal or creatinine clearance > 50 mL/min
* total bilirubin within institutional limits (unless elevated from documented Gilbert's syndrome)
* AST and ALT ≤ 2.5 X institutional upper limit of normal (≤ 5 x institutional upper limit of normal in the presence of liver metastases)
* platelet count ≥ 100,000/µL
* absolute neutrophil count (ANC) ≥ 1500/µL
* Hgb ≥ 9.0 g/dL
* patients with previously treated brain metastases who are not on corticosteroids are eligible
* effective contraceptive method (e.g., intrauterine device, oral contraceptive, or barrier device) must be used during the study by male and female patients of childbearing potential
* ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

* patients who have had immunotherapy, chemotherapy, or radiotherapy within 4 weeks (within 6 weeks for nitrosoureas or mitomycin C) prior to study entry; study entry defined as first day of drug dosing
* patients who have undergone major surgery within 4 weeks prior to study entry
* patients who are receiving another investigational drug
* patients with active CNS metastases or leptomeningeal disease not controlled by prior surgery or radiotherapy
* uncontrolled illness including but not limited to: ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV heart failure), unstable angina pectoris, cardiac arrhythmia, and psychiatric illness that would limit compliance with study requirements
* risk factors for QTc prolongation and/or Torsade de Pointes
* patients with known HIV infection
* concurrent systemic hormonal therapy except: stable LHRH agonist therapy for prostate cancer; hormonal therapy (e.g., megestrol) for appetite stimulation; nasal, ophthalmic, and topical glucocorticoid preparations when appropriate; stable oral glucocorticoid and mineralocorticoid replacement for adrenal insufficiency; or oral contraceptives
* patients who have other medical or psychiatric illness or organ dysfunction which, in the opinion of the Investigator, would either compromise the patient's safety or interfere with the evaluation of the safety of the study agent
* pregnant or lactating women (female patients must have a negative serum pregnancy test within 7 days of study entry)
* patients who have previously received histone deacetylase inhibitors

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Undevia, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- See also: Pharmacyclics — http://www.pharmacyclics.com